CLINICAL TRIAL: NCT00242463
Title: The Efficacy of Anabolic Steroids for the Nutritional Rehabilitation of Critically Ill Patients
Brief Title: Anabolic Steroids for Nutritional Rehabilitation of Critically Ill Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: drug no longer available in canada
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Dr. M. Sharpe, Lawson Health Research Institute
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R-05-390; 11582 (Other: REB)
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Malnutrition; Critical Illness
Keywords: malnutrition; anabolic steroids; intensive care unit; rehabilitation
MeSH Terms: conditions — Malnutrition; Critical Illness | interventions — Nandrolone; Anabolic Androgenic Steroids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- nandrolone (Experimental): Patients receive weekly injections of nandrolone
  Interventions: Drug: Nandrolone (anabolic steroid)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nandrolone (anabolic steroid)
  Arms: nandrolone
Drug: Placebo
  Arms: Placebo

SUMMARY:
This prospective, double-blinded study will determine the feasibility of determining the efficacy of a weekly intramuscular injection of nandrolone (an anabolic steroid) in malnourished ICU patients.The data from this study will also enable us to prepare a future grant proposal with a calculated sample size necessary to demonstrate an improvement in clinical outcome.

DETAILED DESCRIPTION:
Critically ill patients are particularly prone to excessive catabolism using skeletal muscle as the primary substrate as a result of maladaptation to critical illness. Ultimately, critical illness leads to a significant loss of lean body mass (LBM). For example, a 40% loss of LBM is associated with a 100% mortality. Anabolic steroids have been studied and have been shown to improve nutrition in select malnourished patient groups, however, the majority of these studies were not well designed or consisted of small sample sizes.

Our hypothesis is anabolic steroid administration will result in an augmentation of positive nitrogen balance and LBM. This increase in LBM will result in liberation from mechanical ventilation sooner than the placebo group and will result in discharge from the ICU sooner, and as a result, a reduction in morbidity (nosocomial infections) and possibly mortality.

All moderately to severly malnourished ICU patients who have an anticipated stay in ICU > 10 days, will be randomized to receive nandrolone (25 mg-females, 50 mg;males) once weekly for six weeks or placebo. All patients will receive a standard enteral nutritional regimen. Patients will be monitored for assessment of nitrogen balance, lean body mass, and length of time spent on ventilator, in ICU and in HOSP, and incidence of infections.Lean body mass will be measured using a bioimpedance analyzer.

ELIGIBILITY:
Inclusion Criteria:

1. anticipated length of stay in ICU >10 days
2. moderate to severe malnutrition
3. patient tolerating enteral feeds

Exclusion Criteria:

1. age < 18 yrs
2. known allergy to nandrolone
3. women of child bearing age with positive pregnancy test
4. contraindications to intramuscular injections ie anticoagulation
5. renal failure requiring renal replacement therapy
6. patients with breast or prostate cancer -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Nitrogen Balance

SECONDARY OUTCOMES:
Lean body mass
serum prealbumin
length of stay on ventilator, in ICU, in HOSPITAL
infectious complications
outcome (mortality)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Sharpe, MD FRCPC, Principal Investigator — London Health Sciences Centre-UC
Locations (1):
- London Health Sciences Centre-UC, London, Ontario, Canada

REFERENCES:
- [Background] Chang DW, DeSanti L, Demling RH. Anticatabolic and anabolic strategies in critical illness: a review of current treatment modalities. Shock. 1998 Sep;10(3):155-60. doi: 10.1097/00024382-199809000-00001. PMID 9744642
- [Background] Johansen KL, Mulligan K, Schambelan M. Anabolic effects of nandrolone decanoate in patients receiving dialysis: a randomized controlled trial. JAMA. 1999 Apr 14;281(14):1275-81. doi: 10.1001/jama.281.14.1275. PMID 10208142